CLINICAL TRIAL: NCT03483272
Title: MR-flow to Validate Hemodynamic Effect of Terlipressin in Patients With Acute Hepatorenal Syndrome: Can MRI and Echocardiography Predict the Pharmacological Response and Longterm Effect of Terlipressin?
Brief Title: MRI to Assess the Effect of Terlipressin in Patients With Acute Hepatorenal Syndrome (HRS-AKI)
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Flemming Bendtsen, Professor, Hvidovre University Hospital
Other Study IDs: 17001401
Record Dates: First submitted 2018-03-14; First posted 2018-03-30 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Hepato-Renal Syndrome; Portal Hypertension; Acute Kidney Injury; Liver Diseases; Liver Cirrhoses; Cirrhosis Cardiac; Cirrhosis
Keywords: Terlipressin; Pharmacological respons; Magnetic Resonance Imaging; Hemodynamic assessments; Echocardiography; Hepatorenal syndrome - acute kidney injury
MeSH Terms: conditions — Hepatorenal Syndrome; Hypertension, Portal; Acute Kidney Injury; Liver Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard clinical blood tests and pertinent bioactive substances is measured in blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heptorenal syndrome (HRS) is divided into two types. A non-acute kidney injury (NAKI-HRS), which is predominantly related to end-stage disease and a more acute kidney injury (HRS-AKI). HRS-AKI is potentially reversible and develops subsequent to aggravation of a systemic circulatory vasodilatation, that triggers renal vasoconstriction and deteriorates renal perfusion and function. The albumin and terlipressin response is evaluated clinically, routinely for a week and reduces mortality with 23% compared to no treatment. Only 40-50% of the patients with HRS-AKI respond to the treatment with terlipressin.

The treatment of hepatorenal syndrome (HRS-AKI) is aimed at improving blood flow to the kidneys. Flow changes associated to development of HRS have only sparsely been studied and not previously by MR technique and no previous studies have evaluated changes in flow induced by terlipressin. It has been hypothesized that development of HRS is associated to a deterioration in heart function with development of cardiomyopathy, which together with renal vasoconstriction leads to renal failure. Simultaneous MR-assessments of cardiac function and flows (especially the renal flow) in HRS-AKI have not previously been performed.

The aim of the project is to develop new, fast and non-invasive methods to evaluate hemodynamic changes and individual pharmacological terlipressin response in patients with acute hepatorenal syndrome (type HRS-AKI)

We expect a higher increase in renal blood flow in terlipressin-responders compared to terlipressin-non-responders and non-responders will generally have a lower basic renal flow and a decreased cardiac output.

Study design and patients The study design is experimental and includes 30 cirrhotic patients with HRS-AKI. Patients with HRS-AKI are MR scanned before and 17 minutes after their first dose of terlipressin. ECHO is performed before first dose of Terlipressin and is repeated after one of the first doses of terlipressin. Clinically efficacy is defined in accordance to international guidelines at day-7 and 90 days mortality is registered. The screening period and treatments follow international and national guidelines for acute renal failure in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and acute hepatorenal syndrome (HRS-AKI)
* Patient of more than 18 and less than 78 years of age

Exclusion Criteria:

* Patients who are unable to give informed consent
* Patients with absolute contraindication for MRI
* Patients with absolute contraindication for terlipressin
* Pregnant women
* Patient with severe hemodynamic comorbidity

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with cirrhosis and acute kidney injury who meet the criteria for HRS-AKI and needs terlipressin treatment.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Flow (mL/min) in kidney and splanchnic vessels in patients with HRS-AKI and cirrhotic patients without kidney impairment | Baseline (mL/min)
  i) To characterize and compare changes in flow with MR and ECHO in patients with HRS-AKI compared to cirrhotic patients without kidney impairment

SECONDARY OUTCOMES:
Flow changes (mL/min) in HRS-AKI patients with terlipressin non-response vs. response. | Response after 7 days treatment (mL/min)
  To investigate whether flow changes measured with MR and echocardiography induced by a single dose of terlipressin can predict the clinical (7 days) response to terlipressin treatment.
  Full terlipressin response is if creatinine level returns to baseline after 7 days treatment.
  Partial response is a reduction in creatinine of 25% after 7 days terlipressin treatment
Flow changes (mL/min) after terlipressin administration compared to mortality. | 90 days
  To investigate whether flow changes measured with MR and echocardiography induced by a single dose of terlipressin can predict the mortality after 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bendtsen, Study Chair — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Hvidovre University Hospital, Hvidovre, Capital Region
  - Centre of Gastroenterology, Dept. of medicine. Hvidovre University Hospital, Hvidovre

REFERENCES:
- [Derived] Danielsen KV, Hove JD, Nabilou P, Kronborg TM, Wiese S, Siebner HR, Scott R, Francis ST, Aithal GP, Moller S, Bendtsen F. Mapping the hemodynamic effects of terlipressin in patients with hepatorenal syndrome using advanced magnetic resonance imaging. JHEP Rep. 2025 May 10;7(8):101452. doi: 10.1016/j.jhepr.2025.101452. eCollection 2025 Aug. PMID 40677691